CLINICAL TRIAL: NCT01643980
Title: Prevention of Preterm Birth in Pregnant Women at Risk Identified by Ultrasound: Evaluation of Two Treatment Strategies
Acronym: PESAPRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dra.Cristina Martinez Payo (Other)
Responsible Party: Sponsor-Investigator, Dra.Cristina Martinez Payo, Principal Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PESAPRO-2012; 2012-000241-13 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-07-18 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Early Onset of Delivery Before 37 Weeks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal micronized progesterone (Experimental): 200 mg vaginal route per day
  Interventions: Drug: Vaginal micronized progesterone
- Cervical pessary (Active Comparator): Cervical pessary certified by European Conformity (CE0482, MED/CERT ISO 9003/EN 46003;Dr Arabin, lower larger diameter 70 mm, height 30 mm,and upper smaller diameter 32 mm)
  Interventions: Device: Cervical pessary

INTERVENTIONS:
Drug: Vaginal micronized progesterone — 200 mg vaginal route per day
  Arms: Vaginal micronized progesterone
Device: Cervical pessary — Cervical pessary certified by European Conformity (CE0482, MED/CERT ISO 9003/EN 46003;Dr Arabin, lower larger diameter 70 mm, height 30 mm,and upper smaller diameter 32 mm)
  Arms: Cervical pessary

SUMMARY:
The preterm birth is considered as a main problem in the modern obstetrics, being the responsible of greatest of 50% neonatal morbimortality and heavy costs. Despite the significant medical advances, the rate of prematurity has not declined over the past 40 years and even continues to rise in the developed countries. In order to decrease the prematurity is necessary that two premises: to identify the pregnant women at risk of preterm birth, and dispose of useful measures aimed at prolonging the pregnancy and therefore avoid preterm delivery. The investigators propose a clinical trial with the objective to identify effective strategies to reduce the premature birth (34 weeks and earlier) rate in the population of pregnant women at risk for premature birth, which will be identified by ultrasound during the second trimester of their pregnancy.

The investigators intend to compare two accepted strategies: administration of progesterone (vaginally) or the placement of vaginal pessaries. These 2 strategies are affordable, easy to apply, and they present very few maternal-fetal secondary effects.

DETAILED DESCRIPTION:
The preterm birth is considered as a main problem in the modern obstetrics, being the responsible of greatest of 50% neonatal morbimortality and heavy costs. Despite the significant medical advances, the rate of prematurity has not declined over the past 40 years and even continues to rise in the developed countries. In order to decrease the prematurity is necessary that two premises: to identify the pregnant women at risk of preterm birth, and dispose of useful measures aimed at prolonging the pregnancy and therefore avoid preterm delivery. Since 1990, many published articles describe the sonographic measurement of the cervix from the week 16 as method of population screening to detect women at risk. Several studies provide evidence about an inverse relationship between the cervical length and the risk of preterm delivery. For this reason, if there is an effective intervention for patients with cervix short (about < 25mm), made this measure in the middle of the second term, the investigators could reduce the prematurity. Regarding possible therapeutic strategies, recent published data demonstrate the effective of vaginal progesterone and cervical pessary in this population. However, both treatments have never been compared and none of the two strategies are indicated in this population. Therefore it results necessary to compare both treatments in order to establish clinical recommendations. The investigators propose a clinical trial to compare two accepted strategies: administration of progesterone (vaginally) or the placement of vaginal pessaries in order to reduce the premature birth (34 weeks and earlier) rate in the population of pregnant women at risk for premature birth, which will be identified by ultrasound during the second trimester of their pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with short cervix (=< 25 mm) identified by use of routine transvaginal ultrasonography at 19-22 weeks of gestation.
* Single pregnancy
* Women older than 18 year-old
* Women sign informed consent according GCP and local legislation
* Gestational age at randomization between 20+1 and 23+6 weeks.

Exclusion Criteria:

* Major fetal abnormalities
* Major uterine abnormalities
* Placenta praevia during current pregnancy
* Vaginal bleeding or ruptured membranes in the moment of randomization
* Cervical cerclage in situ
* History of cone biopsy
* Allergic to peanuts
* Contraindication for Progesterone usage.
* Active treatment with Progesterone at randomization.
* History of 3 or more premature labor.
* If in the investigator's opinion, there are findings on physical examination, abnormalities in the results of clinical analyzes or other medical factors, social or psycho-social that could negatively influence.
* Women unable to give the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-08; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of spontaneous preterm birth before 34 weeks of gestation | up to 11 weeks (from date of randomization until delivery)

SECONDARY OUTCOMES:
Proportion of spontaneous preterm birth before 37 weeks of gestation | up to 17 weeks (from date of randomization until delivery)
Proportion of Spontaneous preterm birth before 28 weeks of gestation | up to 8 weeks (from date of randomization until delivery)
Rate of premature rupture of membranes before 34 weeks of gestation | up to 11 weeks (from date of randomization until delivery)
Weight at birth | up to 21 weeks (from date of randomization until delivery)
Rate of fetal and neonatal mortality | From date of randomization until the date of delivery, assessed up 21 weeks
Symptomatic vaginal infections during treatment period | From date of randomization until the date of delivery, assessed up 21 weeks
Proportion of participants with adverse events | From date of randomization until the date of delivery, assessed up 21 weeks
Rate of Chorioamnionitis during third term | From date of randomization until the date of delivery, assessed up 21 weeks
Need of admission because of premature labor before 34 weeks of gestation | up to 14 weeks (from date of randomization until delivery)
Rate of neonatal morbidity | From date of randomization until the date of delivery, assessed up 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cruz Melguizo, Dr, Principal Investigator — University Hospital Puerta de Hierro Majadahonda; Cristina Martinez Payo, Dr., Principal Investigator — University Hospital Puerta de Hierro Majadahonda
Locations (27):
- Spain (27):
  - University Hospital San Juan de Alicante, Sant Joan d'Alacant, Alicante
  - University Hospital Quiron Dexeus, Barcelona, Barcelona
  - Igualada Hospital, Igualada, Barcelona
  - Burgos University Hospital, Burgos, Burgos
  - Ciudad Real General University Hospital, Ciudad Real, Ciudad Real
  - Guadalajara General University Hospital, Guadalajara, Guadalajara
  - University Hospital de León, León, León
  - University Hospital Príncipe de Asturias, Alcalá de Henarés, Madrid
  - University Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - University Hospital Madrid Monte Principe, Boadilla del Monte, Madrid
  - University Hospital Fuenlabrada, Fuenlabrada, Madrid
  - University Hospital de Getafe, Getafe, Madrid
  - University Hospital Severo Ochoa, Leganés, Madrid
  - Sanitas La Zarzuela Hospital, Madrid, Madrid
  - University Hospital Ramón y Cajal, Madrid, Madrid
  - Sanitas La Moraleja Hospital, Madrid, Madrid
  - University Hospital Puerta de Hierro, Majadahonda, Madrid
  - University Hospital Rey Juan Carlos I, Móstoles, Madrid
  - University Hospital Mostoles, Móstoles, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Infanta Elena, Valdemoro, Madrid
  - University Hospital Quirón Málaga, Málaga, Málaga
  - Palamos Hospital, Girona, Palamos
  - Hospital Universitario de Donostia, Donostia / San Sebastian, San Sebastian
  - Valladolid Clinic Universitary Hospital, Valladolid, Valladolid
  - University Hospital Rio Hortega, Valladolid, Valladolid
  - University Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Cruz-Melguizo S, San-Frutos L, Martinez-Payo C, Ruiz-Antoran B, Adiego-Burgos B, Campillos-Maza JM, Garcia-Gonzalez C, Martinez-Guisasola J, Perez-Carbajo E, Teulon-Gonzalez M, Avendano-Sola C, Perez-Medina T. Cervical Pessary Compared With Vaginal Progesterone for Preventing Early Preterm Birth: A Randomized Controlled Trial. Obstet Gynecol. 2018 Oct;132(4):907-915. doi: 10.1097/AOG.0000000000002884. PMID 30204689
- [Derived] Cabrera-Garcia L, Cruz-Melguizo S, Ruiz-Antoran B, Torres F, Velasco A, Martinez-Payo C, Avendano-Sola C; PESAPRO trial Group. Evaluation of two treatment strategies for the prevention of preterm birth in women identified as at risk by ultrasound (PESAPRO Trial): study protocol for a randomized controlled trial. Trials. 2015 Sep 25;16:427. doi: 10.1186/s13063-015-0964-y. PMID 26407852